Official Title: Comparison of Efficacy of Rifaximin, Probiotics and LOLA (L-Ornithine L-Aspartate) in Overt Hepatic Encephalopathy: A Randomized, Phase-IV, Lactulose Controlled Clinical Trial.

NCT number: not assigned yet

Date: 25 August 2023

## CONSENT FORM

Title: Comparison of Efficacy of Rifaximin, Probiotics and LOLA (L-Ornithine L-Aspartate) in Overt Hepatic Encephalopathy: A Randomized, Phase-IV, Lactulose Controlled Clinical Trial.

| Name of PI | Qurratulain Jamil |
|---------------------|-------------------|
| Participant name | |
| Screening ID number | |

## STATEMENT OF PERSON GIVING CONSENT:

- 1. I confirm that I have read the information sheet for the study above, or it has been explained to me in a language I am familiar with.
- 2. I have spoken with the doctor to my satisfaction, and I've had the chance to ask any questions I had.
- 3. I understand that my participation is completely voluntary. I have received sufficient information about the research study to decide whether I want to take part.
- 4. I understand that I have the freedom to withdraw at any time, without giving any explanation and that my medical care or legal rights will not be compromised.
- 5. I am aware that I will receive a copy of this consent form and the information sheet to keep for my records.
- 6. I understand that the study staff might look into some of my medical records and I give them permission to do so.
- 7. I am aware that my data will be available to the public with all personal information omitted.
- 8. I agree to a copy of this consent form which includes my personal information being made available to Department of Pharmacy Practice, Faculty of Pharmacy, The Islamia University of Bahawalpur for the purpose of monitoring only.
- 9. I consent to participate in the study mentioned above.

| Name of patient | Date | Signature/ thumbprint or other mark (if unable to sign) |
|---|---|---|
| Name of witness | <br> | <br> |
| (witness if patient is unable | to read or write) | |
| STATEMENT OF PERSON ( | OBTAINING INFORMED CO | NSENT |
| I have provided a detail<br>make an informed decis | _ | search to the participant, including the risks and benefits to |
| <br>Name | <br> | |